CLINICAL TRIAL: NCT05220332
Title: Abundant Living: A Church-based Intervention to Improve Blood Pressure in African Americans
Brief Title: Church-based Intervention to Improve Blood Pressure in African Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Lynch, Associate Professor, Rush University Medical Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18050306
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart to Heart (Experimental)
  Interventions: Behavioral: Heart to Heart
- Money Smart (Active Comparator)
  Interventions: Behavioral: Money Smart

INTERVENTIONS:
Behavioral: Heart to Heart — The Heart to Heart intervention will be delivered at the churches over 6 months. The intervention consists of 12 bible study sessions (45 minutes) led by the Senior Pastor and 24 behavior change small group sessions (90 minutes) led by a trained Rush staff interventionist. These sessions are open to the entire church membership and focus on improving diet and physical well being. A community health worker will provide individualized support to participants with uncontrolled blood pressure who do not reduce their blood pressure by participating in small groups.
  Arms: Heart to Heart
Behavioral: Money Smart — The Money Smart program for adults was developed by the Federal Deposit Insurance Corporation (FDIC). It consists of training modules that cover basic financial topics including deposit and credit services offered by financial institutions, how to obtain and use credit effectively, and the basics of building or repairing credit. This group-based program will be delivered in 14 sessions over 6 months and will be led by a trained instructor.
  Arms: Money Smart

SUMMARY:
This is a 12-month behavioral cluster-randomized trial testing a church-based intervention to reduce blood pressure in African Americans with uncontrolled blood pressure.

ELIGIBILITY:
Inclusion Criteria:

Churches:

* At least 75 members and ability to recruit 15 study participants
* Predominantly African American congregants

Participants:

* Age 18 or older
* Has blood pressure readings with uncontrolled blood pressure, defined as exceeding the blood thresholds for initiation of antihypertensive medication according to the 2017 American College of Cardiology/ American Heart Association (ACC/AHA) guidelines.

  - The thresholds are 140/90 for the general population < 65 years old, and 130/80 for individuals ≥ 65 or with diabetes, chronic kidney disease, or high cardiovascular risk (self-report of prior diagnosis of myocardial infarction, coronary heart disease, stroke or heart failure)
* Attends church (virtually or in-person) at least once per month
* Able to attend weekly Zoom meetings
* Consents and completes all baseline assessments

Exclusion Criteria:

Churches:

• Pastor unwilling to conduct Bible study

Participants:

* Unable to make dietary changes due to lack of control over their food source (i.e., eat meals at shelter, nursing home)
* Has a medical condition that prohibits or severely restricts ability to eat vegetables (i.e., renal disease, Crohn's disease)
* Has a medical condition with an uncertain 6-month prognosis
* Inability to give informed consent (i.e., cognitive impairment, does not speak Englis
* Plans to move within the 6 months following enrollment
* Participated in prior ALIVE intervention
* Member of household participating in another church

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Blood pressure | Measured at baseline and 6 months and 12 months after start of the intervention
  The primary outcome is systolic blood pressure at 6 months post start of the intervention. The Omron digital blood pressure monitor will be utilized to measure blood pressure (Omron Healthcare, Inc., Lake Forest, IL). The participant will sit quietly for >5 minutes, 3 readings will be taken 1-2 minutes apart while seated, and an average of the last 2 readings will be taken to evaluate blood pressure.

SECONDARY OUTCOMES:
Change in Medication adherence | Measured at baseline and 6 months and 15 months after start of the intervention
  Medication adherence will be measured using the 15-item Adherence to Refills and Medications Scale (ARMS). The items are evaluated on a 4-point scale ranging from "none of the time" to "all of the time".
Change in DASH diet adherence | Measured at baseline and 6 months and 15 months after start of the intervention
  Adherence to the Dietary Approaches to Stop Hypertension (DASH) diet will be measured using the food frequency questionnaire developed by Viocare (Princeton, NJ). This 156-item graphical, web-based FFQ queries respondents about usual intakes of 156 food and beverage items over the past three months. It also provides food and nutrient analyses to the research team based on the Nutrition Data System for Research 2018 (NDSR, University of Minnesota, Minneapolis, MN).
Change in Self efficacy | Measured at baseline and 6 months and 15 months after start of the intervention
  Self efficacy will be measured using the Hypertension Self-Care Profile Self-efficacy scale which evaluates self efficacy for 8 common self care recommendations for individuals with hypertension. The items are evaluated on a 4-point scale ranging from "not confident" to "very confident".
Change in Quality of life | Measured at baseline and 6 months and 15 months after start of the intervention
  Quality of life will be measured using the EuroQual (EQ-5D-5L) questionnaire. The measure evaluates the participant's perception of their "health today" with respect to mobility, self-care, usual activities, pain/discomfort, and anxiety depression. The items are evaluated on a 5-point scale ranging from "no problem" in the area to "extreme problem" in the area.
Change in Social support | Measured at baseline and 6 months and 15 months after start of the intervention
  Social support for eating a healthy diet will be measured using a 4-item questionnaire which will evaluate the participant's perception of social support received from family members, friends, church members, and their Pastor. The items are evaluated on a 5-point scale ranging from "never" to "always".
Change in Hypertension knowledge | Measured at baseline and 6 months and 15 months after start of the intervention
  Hypertension knowledge will be evaluated using a 10-item questionnaire adapted from the Hypertension Evaluation of Lifestyle and Management (HELM) Knowledge Scale. Systolic and diastolic blood pressure measurements will be evaluated using the following 4 categories: high, low, normal, and don't know. The frequency with which medication should be taken, lifestyle factors associated with hypertension, and health risks associated with hypertension will also be evaluated.
Change in Nutrition knowledge | Measured at baseline and 6 months and 15 months after start of the intervention
  Nutrition knowledge will be evaluated using an 18-item survey adapted from the International Food Policy Study 2020 - United States Survey. Common foods and food labels are evaluated on a 10-point scale ranging from "not healthy at all" to "extremely healthy".
Change in Barriers to medication use | Measured at baseline and 6 months and 15 months after start of the intervention
  Barriers to medication use will be measured using the 15-item BRIGHT study Barriers to Medication Scale. The scale evaluates different reasons why it is difficult for participants to take medications or to take the medications on time. The items are evaluated on a 5-point scale ranging from "never" to "all the time".

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No